CLINICAL TRIAL: NCT00960596
Title: Preventive Medicine Study of Childhood Atopic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: YungLing Lee / Institute of Preventive Medicine, College of Public Health, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200902042R
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: educational intervention; asthma; Environmental Tobacco Smoke(ETS); children
MeSH Terms: conditions — Asthma | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Health promotion and health education for smoking habits — We provide the education to intervention group.

SUMMARY:
Under environmental intervention programs, to explore the associations between Environmental Tobacco Smoke (ETS) and changes of pulmonary function, cytokines and new-onset asthma between different groups.

DETAILED DESCRIPTION:
Environmental intervention programs:

We will both interview by telephone and mail the health education leaflets, in order to achieve the following aims:

-Smokers living with the children will change where smoking takes place for reducing the children's ETS exposure.

Data collection:

We will contact participants individually to get informed consent before data collection. No matter what intervention, non-intervention or reference group, all participants will test as follows:

* Blood sample collection: We will test the total IgE, specific IgE, cytokines, such as IL-4, IL-13, TNF-α, ECP and EOS.
* Questionnaire collection
* Pulmonary function test

After intervention programs applied, all participants will test pulmonary function, and total IgE, specific IgE and cytokines by blood sample after six months by school approaches. Then, we can compare the pulmonary function, total IgE, specific IgE and cytokines before and after intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Only one smokers living in the same household
* Having smoking exposure during the past 12 months while questionnaire surveying
* Child without smoking habit

Exclusion Criteria:

* None of above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
urine cotinine level | six months, one year

CONTACTS AND LOCATIONS:
Overall Officials: YungLing Lee, Dr., Principal Investigator — Institute of Preventive Medicine, College of Public Health, National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan